CLINICAL TRIAL: NCT05266638
Title: AgeTLIF - Assessing Risk Factors for Radiological Complications After Transforaminal Lumbar Interbody Fusion
Brief Title: Assessing Risk Factors for Radiological Complications After Transforaminal Lumbar Interbody Fusion
Acronym: AgeTLIF
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02227; mu22Netzer
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Lumbar Spine Diseases
Keywords: Posterior Lumbar Interbody Fusion (PLIF); Transforaminal Lumbar Interbody Fusion (TLIF); Implant Failure; Revision Surgery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection (radiological parameters, outcome information) from electronic patient files in hospital data system — Collection of medical data and medical images (MRI, radiographs) of the lumbar spine and pelvis of patients having received TLIF with degenerative spinal diseases from the years 2015-2020 and statistical analysis of the coded data.

SUMMARY:
This retrospective study is to determine whether age is a risk factor for postoperative complications in patients undergoing transforaminal lumbar interbody fusion; specifically whether the risk (odds) of implant failure and the need for revision surgery increases with age.

DETAILED DESCRIPTION:
Spinal fusion is one of the most commonly performed surgical procedures for the treatment of degenerative spinal disease. Interbody fusion with cages reconstructs the anterior column through disc removal, allowing to maintain proper disc height despite weight bearing, while providing firm fixation of the spinal segments. Transforaminal lumbar interbody fusion (TLIF) has fewer complications and less intraoperative bleeding than posterior lumbar interbody fusion (PLIF). Elderly patients are at high risk for perioperative and postoperative complications after lumbar fusion. This retrospective study is to determine whether age is a risk factor for postoperative complications in patients undergoing transforaminal lumbar interbody fusion; specifically whether the risk (odds) of implant failure and the need for revision surgery increases with age.

ELIGIBILITY:
Inclusion Criteria:

* Indications for TLIF surgery (e.g., degenerative disc disease, spondylolisthesis)
* Existing preoperative upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis, sacrum and femoral head
* Existing preoperative MRI of the lumbar region with clear visibility of different fatty infiltration grade and stenosis degree
* Complete follow-up at 3 months and 1 year postoperatively, including clinical and radiographic data

Exclusion Criteria:

* Neuromuscular diseases such as Parkinson's disease or multiple sclerosis according to our records
* Preoperative infection and/or malignancy tumor with involvement of the bony or soft tissue structures of the lumbar spine
* Presence of a documented consent dissent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received TLIF at the age of 55 years or older at the University Hospital Basel between 01.01.2015 and 1.07.2020.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Implant failure | one time assessment at baseline
  Number of Implant failure (screw loosening, cage subsidence, adjacent level alteration/ degeneration, spondylolisthesis degree, kyphosis of the adjacent intervertebral disc space, reduced height of intervertebral disc space) in relationship to age
Number of patients needing revision surgery | one time assessment at baseline
  Number of patients needing revision surgery, in relationship to age

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Netzer, PD Dr. med., Principal Investigator — University Hospital Basel, Clinic for Orthopedics and Traumatology
Locations (1):
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland